CLINICAL TRIAL: NCT07093073
Title: A Single-arm, Open-label Clinical Study Evaluating the Efficacy and Safety of U01 (ssCART-19) in Patients With Relapsed or Refractory B-cell Lymphoma.
Brief Title: Clinical Study of U01（ssCART-19） in Patients With B-Cell Lymphoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Unicar-Therapy Bio-medicine Technology Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: U01
Record Dates: First submitted 2025-07-21; First posted 2025-07-30 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: B Cell Lymphoma
Keywords: CD19; ssCART-19
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- U01(ssCART-19) CAR-T cells (Experimental): CD19-targeted CAR-T cells engineered with an IL-6 silencing element
  Interventions: Drug: ssCART-19

INTERVENTIONS:
Drug: ssCART-19 — Lymphodepletion preconditioning is required prior to CAR-T cell therapy. Lymphodepletion will be performed using a regimen of cyclophosphamide (250-500 mg/m²) and fludarabine (25-30 mg/m²), each administered for 3 consecutive days.

SUMMARY:
This is a single-arm, open-label clinical study evaluating the efficacy and safety of U01 (ssCART-19) in patients with relapsed or refractory B-cell lymphoma.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the efficacy and safety of CD19-targeted CAR-T cells engineered with an IL-6 silencing element in patients with relapsed or refractory B-cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary written informed consent obtained from the participant (or legal guardian) with good compliance expected throughout the study.
2. All of the following conditions must be met:

   1. Age 2-75 years at informed consent; both sexes eligible. For minors (≤18 years), consent must be provided by a parent/legal guardian; minors able to sign must co-sign with their guardian.
   2. Histologically confirmed B-cell lymphoma per the 2024 v3 NCCN Clinical Practice Guidelines in Oncology: B-Cell Lymphomas.
   3. Prior therapy requirements:

      * Failure to achieve PR after first-line therapy, OR relapse within 12 months after first-line therapy; or Relapsed/refractory after second-line therapy (one standard chemo-regimen + one salvage regimen).

   Prior regimens must have included anti-CD20 monoclonal antibody (unless documented CD20-negative tumor) and an anthracycline-containing regimen. In addition, at least one of the following must apply:

   i. Ineligible for autologous hematopoietic stem-cell transplantation (ASCT); ii. Refusal of ASCT; iii. Relapse after ASCT. d) Disease status at screening:

   • Relapse: progression after prior PR or CR.

   • Refractory: i. PD during/after last therapy, or best response ≤SD lasting <6 months; OR ii. Relapse or progression after ASCT (biopsy-proven), including relapse/PD ≤12 months post-ASCT or lack of response (SD/PD) to salvage therapy after ASCT.
3. Tumor tissue (archival or fresh) positive for CD19 by IHC; pathology report within 6 months preferred.
4. ≥1 measurable lesion per Lugano 2014 response criteria.
5. ECOG performance status 0-3.
6. Adequate marrow reserve: ALC ≥0.3 × 10⁹/L; PLT ≥30 × 10⁹/L (transfusion permitted).
7. Adequate organ function:

   • AST ≤3×ULN (≤5×ULN if tumor-related); ALT ≤3×ULN (≤5×ULN if tumor-related);• Total bilirubin ≤2×ULN (≤3×ULN with direct bilirubin ≤1.5×ULN for Gilbert's syndrome);• Serum creatinine ≤1.5×ULN or creatinine clearance ≥60 mL/min (Cockcroft-Gault);• Pulmonary: ≤Grade 1 dyspnea and SpO₂ >91 % on room air;• LVEF ≥50 % by echocardiography;• INR ≤1.5×ULN and APTT ≤1.5×ULN.
8. Women of child-bearing potential: negative serum/urine pregnancy test within 7 days before CAR-T infusion. All participants with reproductive potential must use effective contraception from screening through ≥12 months after CAR-T infusion.
9. Adequate venous access for leukapheresis or repeated phlebotomy, with no contraindications to leukapheresis.
10. Estimated life expectancy >3 months.

Exclusion Criteria:

1. Concurrent malignancy other than the study indication, except for carcinoma in situ or any malignancy with a disease-free interval ≥3 years.
2. Presence of any of the following:• Positive HBe-Ab and/or HBc-Ab with HBV-DNA above the lower limit of quantification;• Positive HCV-Ab with HCV-RNA above the lower limit of quantification;• Positive Treponema pallidum antibody (TP-Ab);• Positive HIV antibody.
3. Active bacterial, fungal, viral, mycoplasmal, or other infection deemed uncontrollable by the investigator.
4. History or current clinically significant CNS disorder unrelated to lymphoma-e.g., seizure disorder, cerebral ischemia/hemorrhage, dementia, cerebellar disease, or any CNS autoimmune disease-that the investigator considers uncontrolled.
5. Within 12 months before informed consent: percutaneous coronary intervention (angioplasty or stent placement), NYHA Class III-IV congestive heart failure, myocardial infarction, unstable angina, or other clinically significant cardiac history judged by the investigator; or QTc >480 ms (Fridericia correction) or LVEF <50 % by echocardiography at screening.
6. Known primary immunodeficiency.
7. History of severe immediate hypersensitivity to any study drug.
8. Receipt of any live vaccine within 6 weeks before screening.
9. Pregnant or breastfeeding women.
10. Active autoimmune disease requiring systemic immunosuppressive therapy.
11. Participation in any other interventional clinical trial within 30 days before signing informed consent.
12. Any condition that, in the investigator's opinion, renders the subject unsuitable for study participation.

Ages: 2 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01-23 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse events after U01 CAR-T cells infusion [Safety and Tolerability] | 28 days post administration of ssCART-19
  An assessment of severity grade will be made according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE)
Objective Response Rate (ORR), as assessed by Investigators | 2 years post CAR T cell infusion
  The Objective Response Rate (ORR) is the percentage of participants who achieved a best overall response of Complete Remission (CR) or Partial Remission(PR)
Duration of response (DOR) | 2 years post CAR T cell infusion
  Duration of response (DOR) is defined as the time from the first documented objective response to the first documented disease progression or death.
Overall survival (OS) | 2 years post CAR T cell infusion
  Overall Survival (OS) was defined as the time from the date of first infusion of U01 to the date of death due to any cause.
Progression-free survival (PFS) | 2 years post CAR T cell infusion
  Progression-free survival (PFS) was defined as the time from the date of infusion to the earliest date of the first objective documentation of progressive disease (PD) or death due to any cause.

SECONDARY OUTCOMES:
Pharmacokinetics of ssCART-19 | 2 years post CAR T cell infusion
  Time at the maximal concentration(Tmax)
Pharmacokinetics of ssCART-19 | 2 years post CAR T cell infusion
  Area under the concentration-time curve(AUC)
Pharmacokinetics of ssCART-19 | 2 years post CAR T cell infusion
  The maximal concentration of peripheral blood (Cmax)
Pharmacodynamics of ssCART-19 | 2 years post CAR T cell infusion
  Concentration levels of CAR-T-related serum cytokines such as IL-6, IFN γ, ferritin and CRP at each time point

CONTACTS AND LOCATIONS:
Overall Officials: Wenjun Zhang, Ph.D., Principal Investigator — Tongji Hospital
Locations (3):
- China (3):
  - Hebei Yanda Lu Daopei Hospital, Hebei
  - Tongji Hospital of Tongji University, Shanghai
  - Tianjin First Central Hospital, Tianjin